CLINICAL TRIAL: NCT05648240
Title: Proof-of-concept Study of Blood Markers of Tumor Dissemination in Patients With Versus Without Intestinal Polyps
Acronym: EARDIS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2022-1/JFB01
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Cancer; Neoplasm Metastasis; Disseminated Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood collected at time of colonoscopy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with polyps
  Interventions: Other: Blood test
- Patients without polyps
  Interventions: Other: Blood test

INTERVENTIONS:
Other: Blood test — Venous blood samples taken at the moment of colonoscopy to test for biomarkers

SUMMARY:
The study authors hypothesize that in patients with intestinal polyps, tumor cells could disseminate and circulating factors could be secreted by the polyp. These two parameters could become biomarkers to refine the follow-up of patients and to establish targeted therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patient to be examined by colonoscopy
* The patient must be a member or beneficiary of a health insurance plan

Exclusion Criteria:

* The subject is participating in a category 1 interventional study, or is in a period of exclusion determined by a previous study
* The subject signals their opposition to participate in the study
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Patient pregnant or breastfeeding
* History of proven cancerous disease
* Patient followed for a chronic inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for colonoscopy in the Hepato-Gastro-Enterology Department of the University Hospital of Nîmes. Patients with a family history of colorectal cancer and aged over 50 years, with a positive Fecal Immunological Test, with bleeding, with abdominal pain or with unexplained anemia are all likely to undergo colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2026-02-04 (Actual); Study Completion 2026-02-04 (Actual)

PRIMARY OUTCOMES:
Dissemination of circulating tumor cells in blood samples from patients with intestinal polyps compared to patients without polyps | Day 0
  Number of disseminated circulating tumor cells found on the ANGLE Parsortix™ system

SECONDARY OUTCOMES:
Concentration of Macrophage Colony Stimulating Factor (M-CSF) in the blood samples between groups | Day 0
  ng/mL, measured by Enzyme-Linked ImmunoSorbent Assay
Concentration of Granulocyte Macrophage Colony Stimulating Factor (GM-CSF) in the blood samples between groups. | Day 0
  ng/mL, measured by Enzyme-Linked ImmunoSorbent Assay
Concentration of Chemokine ligand 2 (CCL-2) in the blood samples between groups. | Day 0
  ng/mL, measured by Enzyme-Linked ImmunoSorbent Assay
Concentration of keratinocyte-derived cytokine (CXCL-1) in the blood samples between groups | Day 0
  ng/mL, measured by Enzyme-Linked ImmunoSorbent Assay
Concentration of Tissue Inhibitor of Metalloproteinase 1 (TIMP-1) in the blood samples between groups | Day 0
  ng/mL, measured by Enzyme-Linked ImmunoSorbent Assay
Concentration of Stromal cell-Derived Factor 1 (SDF-1) in the blood samples between groups | Day 0
  ng/mL, measured by Enzyme-Linked ImmunoSorbent Assay
Anti-aggregant therapy according to presence of circulating tumor cells, cytokine presence and presence of polyp | Day 0
  Yes/no
Anti-coagulant therapy according to presence of circulating tumor cells, cytokine presence and presence of polyp | Day 0
  Yes/no
Known intestinal pathology according to presence of circulating tumor cells, cytokine presence and presence of polyp | Day 0
  Yes/no
Reason for screening colonoscopy according to presence of circulating tumor cells, cytokine presence and presence of polyp | Day 0
  Fecal immunochemical test positive / Personal history of colonic adenoma / Family history of colonic adenoma / Personal history of colorectal cancer / Family history of colorectal cancer / Rectal symptoms
Screening colonoscopy operator (inter-operator tumor detection rate) according to presence of circulating tumor cells, cytokine presence and presence of polyp | Day 0
Quality of the preparation according to presence of circulating tumor cells, cytokine presence and presence of polyp | Day 0
  Boston classification: ranked from 0 to 3 for each colonic segment explored
Caecal intubation rate according to presence of circulating tumor cells, cytokine presence and presence of polyp | Day 0
  classed as complete colonoscopy after visualization of the caecal floor
Per-surgical complications according to presence of circulating tumor cells, cytokine presence and presence of polyp | Day 0
  Post-polypectomy bleeding / Perforation / Incomplete colonoscopy / No complications
Total number of colonic adenomas visualized according to presence of circulating tumor cells, cytokine presence and presence of polyp | Day 0
  Number
Total number of histologically validated resected colonic adenomas according to presence of circulating tumor cells, cytokine presence and presence of polyp | Day 0
  Number
Size of resected adenomas according to presence of circulating tumor cells, cytokine presence and presence of polyp | Day 0
  < 5mm / 5 - 10mm / > 10mm
Location of resected adenomas according to presence of circulating tumor cells, cytokine presence and presence of polyp | Day 0
  Rectum / Sigmoid / Left Colon / Transverse Colon / Right Colon / Caecum
Morphology of resected adenomas according to presence of circulating tumor cells, cytokine presence and presence of polyp | Day 0
  Paris classification: 0-Is / 0-Ip / 0-IIa / 0-IIb / 0-IIc / 0-III
Method of resected adenomas according to presence of circulating tumor cells, cytokine presence and presence of polyp | Day 0
  Biopsy forceps / Cold loop / Diathermic loop / Mucosectomy / Unresected (Suspected Cancer, Unresectable in ambulatory)
Recovery of the adenoma after resection according to presence of circulating tumor cells, cytokine presence and presence of polyp | Day 0
  Yes/no
Histology of resected adenomas according to presence of circulating tumor cells, cytokine presence and presence of polyp | Day 0
  Vienna classification: Nonspecific (Food Residue, Normal Mucosa or Colonic Fold) / Adenoma in Low Grade Dysplasia / Adenoma in High Grade Dysplasia / Cancer - Transformed Adenoma / Scalloped Adenoma / Hyperplastic Polyp.
Location of resected adenomas according to presence of circulating tumor cells, cytokine presence and membrane marker expression | Day 0
  Rectum / Sigmoid / Left Colon / Transverse Colon / Right Colon / Caecum

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François BOURGAUX, Principal Investigator — CHU de Nimes
Locations (1):
- CHU de Nîmes, Nîmes, France